CLINICAL TRIAL: NCT00201578
Title: Case Control Study of Non Viral Hepatitis Relating to Herbal Drug Use in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701120
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2005-01

CONDITIONS: Acute Hepatitis
Keywords: Herbal Drugs; Alternative medicine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The use of traditional Chinese herbal medicine and various forms of alternative medicine to maintain health among the Chinese ethnic group has had a long history and has been deeply rooted in the Chinese way of living for centuries. It has been a general belief that these therapies consist of "natural" substances and are less toxic than their western synthetic drug counterparts. However, recent reports of side effects of systemic traditional Chinese medicine, including hypersensitivity, hepatotoxicity, neurotoxicity, cardiovascular toxicity, renal failure, and contact dermatitis, have been increasing.

Since there is a high prevalence in the usage of traditional Chinese herbal medicine in Taiwan, this study examines the frequency of patients using herbal medicine whose initial diagnosis in the emergency department (ED) is acute non viral hepatitis. We, the researchers at National Taiwan University Hospital, then correlate if the cause of hepatitis is related to the use of these herbal drugs by taking a detailed history of medication or herbs used and by verifying the contents by chemical analysis of the "medications" used. To our knowledge, this is the first study in examining the relationship between non viral hepatitis and the use of herbal drugs prior to arriving at the ED. We expect to prove adverse effects of these substances, especially hepatitis, is the cause for requiring emergency care.

Our study design is a prospective, density sampling case control study in which one hundred patients with non viral hepatitis will be recruited as our case. We use a questionnaire designed by the investigator in the survey of demographic background, education, and income status of the cases, as well as the frequency of use of the drug, total dosage used, where the drug was purchased, what the drug is used for, and whether they know of any adverse effect that the drug might have. If they had taken the drug within three months prior to this emergency visit, then they are asked to bring the drug in for examination. Examination of the drug includes the use of high performance liquid chromatography (HPLC) and if necessary, inductively coupled plasma mass spectrometry (ICP mass). In contrast, our control group consists of subjects that are admitted to the ED due to trauma or fracture. For each case, they are matched with two subjects in the control group in both gender and age. They should also arrive within two days after the arrival of the case. All cases and controls are screened for viral hepatitis and serology must be negative before entering the study. The questionnaire is given to both groups. If more than one control is eligible to enter the study, then the control is chosen by a random draw in a hat. After this use of density sampling, we collect the data and logistic regression is used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal liver function test
* Hepatitis other than viral induced

Exclusion Criteria:

* Under age 18 years old
* Viral hepatitis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jung D Wang, Study Director — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan